CLINICAL TRIAL: NCT06020040
Title: The Relationship Between Bone Particles Sizes and the Stability of Soft and Hard Tissue in Aesthetic Area ：3-year Prospective Intervention Clinical Study
Brief Title: Bone Particles Sizes and the Stability of Soft and Hard Tissue in Aesthetic Area
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022（061）
Record Dates: First submitted 2022-05-17; First posted 2023-08-31 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-08

CONDITIONS: Implant Site Reaction
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: The researchers prospectively and continuously recruited subjects who underwent implant therapy with xenogeneic bone graft material in the Oral Implantation Center of the Stomatology Hospital Affiliated to Zhejiang University School of Medicine, and all subjects who signed written informed consent were divided into 2 groups (large bone particles and small bone particles) through a table of random numbers.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study takes a single-blind method. During research process, the researchers cannot avoid knowing the type of abutment used by the subjects during the clinical examination and operation, so the subjects can only be single-blinded. The clinical examination data will be measured and averaged by two independent clinicians. The data will be analyzed by a third person.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large Bone Particles (Experimental): The size of the bone particles that will be used for GBR is 1-2mm.
  Interventions: Device: Heterograft
- Small Bone Particles (Experimental): The size of the bone particles that will be used for GBR is 0.25-1mm.
  Interventions: Device: Heterograft

INTERVENTIONS:
Device: Heterograft — Heterograft (Geistlich, Gegreen, Heal-All) will be used to repair bone defect in the esthetic area of the anterior teeth with simultaneous implant placement. According to the bone particle size, it can be divided into large bone particles(1-2mm) and small bone particles(0.25-1mm).

SUMMARY:
After implant restoration, the surrounding tissue, including the gingiva and alveolar bone, will inevitably reconstruct. The study found that gingival recession was easy to occur in the aesthetic area of upper anterior teeth within 1 year after implantation, which was mainly due to the absorption of labial alveolar bone. In order to avoid absorption, the thickness of the labial bone plate should not be less than 2mm, which is difficult to achieve in the anterior tooth area. Therefore, guided bone regeneration (GBR) should be performed in the implant area, which can provide more than 5mm bone increment in the vertical and horizontal positions with long-term stability, being beneficial for the maintenance of the buccal contour and the stability of the soft and hard tissues in the aesthetic area.

In this study, the inorganic bone matrix extracted from bovine bone (Geistlich, Gegreen, Haiao, etc.) was used for GBR in the area with insufficient bone volume in the anterior dental implant area. The commercially available xenogeneic bone graft substitutes can be divided into large particles (1-2mm) and small particles (0.25-1mm) according to the particle size. Previous studies have found that in 6 months after implantation, the change of vertical bone height around the implant (i.e. the height from the top of alveolar ridge to the shoulder of the implant) is related to the particle size of bone powder, and large particles of bone powder may have better performance in maintaining the vertical bone height due to the following reasons:

1. Large bone particles may show better mechanical properties and better mechanical compression resistance.
2. Large bone particles may show more reasonable pore size and porosity, which may provide better environment for the growth of new bone.
3. Large bone particles may achieve more reasonable and balanced bone remodeling. However, the effect of bone particle sizes on the maintenance of soft and hard tissue around the bone graft area is still inconclusive. Thus, the purpose of this study is to compare the effects of large and small bone particle sizes on the stability of soft and hard tissues around the bone graft area within 3 years after implant restoration in the anterior tooth area.

DETAILED DESCRIPTION:
Research Purpose: To compare the effects of large and small bone particle sizes on the stability of soft and hard tissues around the GBR area within 3 years in the esthetics area of anterior tooth.

Research Design and Methods:

1. Type of study design: prospective intervention single-center randomized clinical trial.
2. Study period: 3 years, from the date of ethics approval to December 2025.
3. This study takes a single-blind method. During research process, the researchers can't avoid knowing the type of abutment used by the subjects during the clinical examination and operation, so the subjects can only be single-blinded.
4. Measures to control bias:

1) Selection bias control: the random number table method was used for grouping, and the blind method was strictly followed in the research process. During the recruiting period, researchers need to be fully informed of the subjects to improve their understanding and compliance with the test. At least two or more contact information should be left in case of minimizing the missed follow-up, and we can contact the subjects in emergency.

2) Control of information bias: rigorous design of case report form, setting up two researchers to collect data independently and try to collect the data of objective indicators, conduct regular researcher training and unify the evaluation criteria.

3) Confounding bias control: improve the research design, control the grouping of single variables, and adopt reasonable statistical analysis methods.

5. When recruit subjects, we will strictly follow the exclusion and inclusion criteria. When subject who meets the following withdrawal criteria, we will terminate the experiment :

1. Implant complications during the study, including but not limited to peri-implantitis and implant fracture, which resulting in implant failure
2. Subjects with poor compliance, unable to review regularly, and do not pay attention to oral hygiene maintenance in daily life
3. Subjects voluntarily asked to withdraw from the study

6. Design plan and specific arrangements: Subjects are expected to participate in clinical trials for 3 years, and need to complete follow-up. Complete preoperative examinations and records will be carried out before surgery, such as gender, age, implant position, smoking, gingival biotype, keratinized gingival width and so on. Imaging examinations, including parallel projection X-rays and CBCT, are required on the day of surgery, 6 months after surgery, 1 year，2 years and 3 years after implant restoration. Gingival tissue information collection (such as mesial and distal gingival papilla, soft tissue color, texture, level and contour, and alveolar ridge) on the day of completion of implant restoration, and 1-year, 2 years and 3 years after implant restoration for Pink Esthetic Score (PES) .

7. Trial suspension criteria: According to the clinical trial protocol:

1. Controllable adverse events occur, or safety problems are found, which can be reasonably controlled by improving the research design or means. Suspend and adjust clinical trial protocols in a timely manner.
2. Some subjects could not avoid the influence of specific risks, so the trial was suspended in time and susceptible subjects were excluded.
3. The data obtained are extremely statistically significant. Apply for an interim analysis.

8. Criteria for termination of the trial:

1. There are serious adverse events, and the adverse events are likely to be related to the intervention in the trial.
2. External information (such as other high-quality research or evidence) proves that the intervention is ineffective or effective, and the current clinical trial is not necessary to continue.
3. According to the planned interim analysis to achieve the expected difference in efficacy, if it has been observed that the intervention program of the experimental group is significantly better than that of the control group.

9. The clinical observations, clinical examination values, imaging measurements, and clinical scale scores generated by the investigator's examination in this study, and original records were made. The source data record shall indicate the record time, record source and recorder.

10. Sample size calculation: In this study, we use horizontal thickness of the labial bone plate as the primary measurement indicator. To the best of our knowledge, no other studies have evaluated the effect of DBBM particle size on LRA outcomes. We will refer to the results of Basma et al., who conducted an LRA study using allografts, to estimate the required sample size. According to previous research, the alveolar bone width increase was 5.1 ± 1.7 mm in the large particle group and 3.1 ± 1.7 mm in the small particle group, resulting in an effect size of 0.925. Using the G*Power software, with a two-tailed t-test, α = 0.05, (1 - β) = 0.85, a case attrition rate of 10%, and an equal group size ratio of 1:1, a total of 50 patients is required.

11. 1) The clinical examination data were measured and averaged by two independent clinicians, recorded in the case collection form, and analyzed by a third person using spss 19.0 statistical software to evaluate whether there were statistical differences. The imaging data were called and analyzed by submitting an application to the Affiliated Stomatology Hospital of Zhejiang University School of Medicine. During the process, the patient's real name was hidden, and the data quality assurance management was carried out according to the following requirements: Exclude all missing data, unused data and illogical data.

2) Screening and sorting out the test data that meet the inclusion criteria, forming a data set of observational safety and various clinical effects and conducting statistical analysis.

3) Modification procedure for deviation from the original statistical analysis plan: submit a deviation report form to the ethics committee. In addition to the deviation statement, the table shows the frequency of each type of deviation and its impact on the research results. Behavior is explained and there are actions taken for deviations from the plan.

4) All records related to the identity of the subjects are kept confidential, and these materials will not be disclosed to the public outside the scope permitted by relevant laws and/or regulations.

12. Statistic analysis: For the collected measurement data, if there is normal distribution data with roughly equal variance, the parameter method (t-test) is used, otherwise, a nonparametric test (Mann-Whitney u test) was used. For the collected counting data (the score of soft tissue around the implant), we used chi-square test.

13. Informed consent:

1. This study will be conducted by the research doctor in the Oral Implantation Center of Zhejiang University Affiliated Stomatology Hospital,and the subjects will be informed and informed consent will be obtained before surgery.
2. The informed consent process conforms to the principles of complete notification, full understanding, and independent choice; the expression of informed consent is easy to understand and conforms to the level of understanding of the subject group.
3. This study does not involve vulnerable groups and all subjects will sign the informed consent form by themselves.

14. Adverse event reporting:This study did not include measures and interventions other than routine clinical treatment, and had no other adverse effects on the subjects.

In the event of an adverse event, we will report it as follows:

1. Various adverse events: Take timely measures to deal with them and record them in the case report form.
2. Serious adverse events (SAE): take measures to deal with them timely, and record in a case report form, stop the trial at the decision of the investigator, immediately report to the ethics committee, drug clinical trial institutions and sponsors, and report to national and provincial food within 24 hours Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years old and above
* 2) Patients with missing maxillary anterior teeth and insufficient horizontal bone mass of alveolar ridge who indeed need GBR
* 3) One-wall or two-wall bone defects
* 4) There is no infection and tooth extraction residue at the implant site
* 5) Simultaneous implant placement
* 6) Subjects who voluntarily join the test cohort and sign the informed consent

Exclusion Criteria:

* 1) Severe periodontitis or uncontrolled periodontitis
* 2) History of head and neck radiotherapy
* 3) History of bisphosphonate administration and injection
* 4) Uncontrolled severe systemic diseases
* 5) Patients with heavy smoking
* 6) Onlay bone graft is needed for bone resorption
* 7) Three-wall or four-wall bone defects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The labial horizontal alveolar bone thickness | pre-surgery, immediately post-surgery, 6 months after operation, 1/2/3-year after implant restoration
  Horizontal bone thickness of implant shoulder, 2mm below the shoulder, 4mm below the shoulder, and 6mm below the shoulder.
The change of Pink esthetic score (PES) from baseline | The day of completion of implant restoration, 0.5/1/2/3-year after implant restoration
  Gingival tissue information collection include mesial and distal gingival papilla, soft tissue color, texture, level and contour, and alveolar ridge. The minimum value is 0, and the maximum value is 14, the higher scores mean a better outcome.

SECONDARY OUTCOMES:
The change of Vertical facial alveolar bone level (VFBL) from baseline | The operation day, 6 months after operation, 1/2/3-year after implant restoration
  The distance from implant shoulder to the highest point of middle facial bone plate

CONTACTS AND LOCATIONS:
Overall Officials: Li Weida, Principal Investigator — Stomatological Hospital Affiliated to Zhejiang University School of Medicine
Locations (1):
- The Stomatologic Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Gao J, Sheng M, Qi W, Jin J, He F. Facial alveolar bone alterations and gray value changes based on cone beam computed tomography around maxillary anterior implants: A clinical retrospective study of 1-3 years. Clin Oral Implants Res. 2020 May;31(5):476-487. doi: 10.1111/clr.13583. Epub 2020 Feb 12. PMID 31990412
- [Background] Kheur MG, Kheur S, Lakha T, Jambhekar S, Le B, Jain V. Does Graft Particle Type and Size Affect Ridge Dimensional Changes After Alveolar Ridge Split Procedure? J Oral Maxillofac Surg. 2018 Apr;76(4):761-769. doi: 10.1016/j.joms.2017.11.002. Epub 2017 Dec 2. PMID 29202263